CLINICAL TRIAL: NCT04434482
Title: A Phase Ib/II, Open-Label, Multi-Center, Dose Escalation and Expansion Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of IMP4297 in Combination With Temozolomide in Patients With Advanced Solid Tumors and Small Cell Lung Cancer
Brief Title: IMP4297 in Combination With Temozolomide in Patients With Advanced Solid Tumors and Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Impact Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMP4297-106
Record Dates: First submitted 2020-06-14; First posted 2020-06-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumours; Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — senaparib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IMP4297(senaparib) and temozolomide (Experimental): IMP4297 and temozolomide
  Interventions: Drug: IMP4297(senaparib)

INTERVENTIONS:
Drug: IMP4297(senaparib) — The dose levels will be escalated following a modified 3+3 dose escalation scheme.
  Other Names: temozolomide

SUMMARY:
This is an open-label, multi-center, dose-escalation and dose-expansion phase I study to evaluate the safety, tolerability, PK characteristics and anti-tumor activity of PARP inhibitor IMP4297 and temozolomide combination therapy in patients with advanced solid tumors and with ES-SCLC who develops disease progression after 1L platinum-based regimen.

DETAILED DESCRIPTION:
This study will be conducted in two parts. Part I of the study will be dose escalation evaluation to determine the MTD and/or recommended phase 2 dose（RP2D） of IMP4297 in combination with temozolomide. Part II of the study will be conducted in two expansion cohorts (sensitive ES-SCLC cohort and resistant ES-SCLC cohort) to further evaluate the anti-tumor activity, safety and tolerability of this regimen in ES-SCLC patients.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must voluntarily participate in this clinical study and be willing and able to provide written informed consent/assent for the trial.
2. Age ≥ 18 years old on the day of signing informed consent form (ICF), males or females
3. Patient population:

   1. In Part I: The patient must have histologically or cytologically confirmed advanced solid tumor that is refractory to standard treatment or for which no standard treatment exists, including but not limited to triple-negative breast cancer (TNBC), SCLC, ovarian cancer (OC) and metastatic castration-resistant prostate cancer (mCRPC).
   2. In Part II: The patients must be histologically or cytologically confirmed ES-SCLC with disease progression after one and only one course of 1L standard platinum-based therapy. Anti-PD-1 or anti-PD-L1 antibody therapy is acceptable as long as it's part of the 1L treatment. Including platinum sensitive and platinum resistant patients. Platinum sensitive is defined as the relapse-free interval exceeds 90 days after treatment with platinum doublets is completed; The platinum resistant represents disease relapses within 90 days of treatment completion during a chemotherapy-free interval (CFI).
   3. In Part I: Patients have an ECOG performance status of 0 to 1.
   4. In Part II: Patients have an ECOG performance status of 0 to 2.
   5. Patients have a life expectancy of ≥12 weeks.
   6. In Part II: patients have at least 1 measurable lesion per RECIST v1.1, including a previously irradiated lesion if has progressed since radiotherapy, that can be accurately measured at baseline which is suitable for accurate repeated measurements
4. Patients have adequate organ function, as indicated by the following laboratory values (had not received blood transfusion, apheresis infusion, erythropoietin, granulocyte colony-stimulating factor, and other relevant medical support within 28 days before the administration of the IPs
5. Female patients should meet at least 1 of the following criteria before they can participate in the study:

   * Females who have no childbearing potential (i.e., physiologically incapable of pregnancy), including those who have undergone hysterectomy, bilateral oophorectomy, or bilateral salpingectomy.
   * Post-menopausal (total cessation of menses for ≥1 year).
   * For those with childbearing potential, they should have a negative serum pregnancy test during the screening period (within 7 days prior to the first dose of the IPs), should not be in lactation, and willing to take effective contraceptive measures throughout the study period, from study entry up to 6 months after the last dose of the IP(s).
6. Male patients are eligible to participate in the study if they have undergone vasectomy or agree to use effective methods of contraception from study entry up to 6 months after the last dose of the IP(s).

Exclusion Criteria:

1. Patients with primary tumor in central nervous system (CNS) and active or untreated central CNS metastases and/or carcinomatous meningitis should be excluded. Patients with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks and, have no evidence of new or enlarging brain metastases and no requirements for corticosteroids 14 days prior to dosing with IPs.
2. Patients with serious acute and chronic infections, including:

   * Patients with an uncontrolled acute infection, or an active infection requiring systemic treatment, or patients who have received systemic antibiotics within 2 weeks prior to the first dose of the IPs; prophylaxis use of systemic antibiotics treatment for upper tract infection is allowed as long as no violation with the requirement in Section 6.5 Concomitant Therapy.
   * Patients who have a known history of human immunodeficiency virus (HIV) infection and/or acquired immunodeficiency syndrome or positive HIV testing should undergo CD4+ T-cell test during the screening period. Patients with CD4+ T-cell counts < 350 cells/uL are ineligible for enrollment. Patients with unknown HIV infection status who are unwilling to undergo HIV testing should not be enrolled in the study;
   * Patients who have known active hepatitis B or C. To be included in the study, patients with hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV) antibody positive test results during screening must be further tested for hepatitis B virus (HBV) DNA titer (excluding patients with a DNA titer of more than 2500 copies [cps]/mL or 500 IU/mL) and HCV RNA (excluding patients with an HCV RNA concentration exceeding the lower detection limit of the assay) to exclude active hepatitis B or hepatitis C infection requiring treatment. Hepatitis B virus carriers, patients with stable hepatitis B infection after drug treatment (DNA titer not exceeding 2500 copies [cps]/mL or 500 IU/mL) and hepatitis C infected patients who received treatment and achieved sustained virologic response for at least 12 weeks can be enrolled.
   * Note: If the lower detection limit of the HBV DNA assay in the study centers is higher than 2500 copies [cps]/mL or 500 IU/mL, the patients in the study center with an HBV DNA assay result lower than the lower detection limit of the assay can be enrolled.
   * Active tuberculosis
3. Patients who have previously received PARP inhibitors.
4. Patients who have received strong CYP3A4 inhibitors or inducers prior to the first dose of the IPs (the patient can be enrolled if the elution period prior to the first dose of the IPs is ≥5 half-lives), or patients who need to continue receiving these medications during the study period.
5. Patients who have received a live-virus vaccination within 28 days of the planned start of study.
6. Patients who have participated a study of an investigational agent and received study therapy or used an investigational device within 28 days of the first dose of treatment.
7. Patients have not recovered (i.e., to ≤Grade 1 or to baseline, as evaluated by NCI-CTCAE v5.0) from cytotoxic therapy-induced AEs, except for alopecia.
8. Patients who have received anti-cancer chemotherapy, endocrine therapy, herbal/alternative therapies (including Chinese herbal or Chinese medicine or proprietary Chinese medicine), or other anti-cancer systemic treatment (except anti-cancer antibody) within 5 half-lives or 14 days, whichever is longer prior to the first dose of the IPs. Patients who have received anti-cancer antibody within 28 days prior to the first dose of the IPs.
9. Patients who have undergone a major surgery within 28 days prior to the study treatment, or have undergone a radical radiotherapy, or have undergone a palliative radiotherapy within 14 days prior to the study treatment, or have used a radioactive drug (Strontium, Samarium, etc.) within 56 days prior to the study treatment.
10. In Part II of the study, patients who have other malignancies within 2 years prior to the first dose of the IPs will be excluded. except for radically treated locally curable malignant tumors, such as basal or squamous cell skin cancer, superficial bladder cancer, or prostate, cervical or breast carcinoma in situ.
11. Patients with uncontrolled pleural effusion, pericardial effusion or ascites requiring recurrent drainage procedures (once monthly or more frequently). Please contact medical monitor if any further discussion or clarification is needed.
12. Patients with a history of seizures.
13. Patients with a previously documented diagnosis of myelodysplastic syndrome (MDS).
14. Patients who have major cardiovascular diseases (such as congestive heart failure, unstable angina, atrial fibrillation, arrhythmia); patients who have acute myocardial infarction, unstable angina, stroke, or transient ischemic attack within 6 months prior to the first dose of the IPs; patients who have congestive heart failure (≥New York Heart Association [NYHA] Classification Class II); patients who have severe arrhythmia requiring medication (including QT interval [QTc] prolongation corrected by the Fridericia's formula [QTcF] of more than 480 msec, pacemaker installation, and previous diagnosis of congenital long QT syndrome).
15. Patients who are unable to swallow capsules. Patients have gastrointestinal illnesses that may affect the absorption of oral medication IMP4297 and temozolomide.
16. Patients with a known hypersensitivity to IMP4297, temozolomide or any of the excipients of the products.
17. Patients who have received transplantation including patients with previous allogeneic bone marrow transplant.
18. Patients known to have a history of alcoholism or drug abuse.
19. The investigator believes that the patient's underlying disease may put the patient at risk in IP administration or may affect the evaluation of toxicity events or AEs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Part I: Dose Escalation safety and tolerability | From signing ICF until safety follow-up
  TEAEs, vital signs, physical examinations, electrocardiogram (ECG), laboratory tests (including serum chemistry, hematology, and urinalysis, coagulation), etc.
Part I: Dose Escalation MTD | from the initiation of study drugs until the end of dose escalation phase(approximately 1 year)
  the maximum tolerated dose:the highest dose level at which <1/3 patients experience DLT
Part I: Dose Escalation RP2D | from the initiation of study drugs until the end of dose escalation phase(approximately 1 year)
  the recommended phase 2 dose
Part II: Dose Expansion Overall Response Rate (ORR) | from the initiation of study drugs until documented disease progression, withdrawal of consent, loss to follow-up, death, initiation of new anti-cancer treatment or termination of study, which occurs first.
  the percentage of patients who had a best response rating of CR and PR which was maintained ≥4 weeks from the first manifestation of that rating.

SECONDARY OUTCOMES:
Part I: Dose Escalation plasma PK profile of IMP4297 and temozolomide | Cycle 1 Day 1, Cycle 1 Day 15,Cycle 2 Day 1,Any cycle after cycle 2,unscheduled visit
  To characterize the plasma PK profile of IMP4297 and temozolomide via population PK (popPK) modeling
Part I: Dose Escalation anti-tumor activity | from the initiation of study drugs until documented disease progression, withdrawal of consent, loss to follow-up, death, initiation of new anti-cancer treatment or termination of study
  Progression-free survival (PFS),Duration of response (DoR),Disease control rate (DCR)
Part I: Dose Escalation,effect of IMP4297 on QT interval | Cycle 1 Day 1,Cycle 1 Day 15,Cycle 2 Day 1,CnD1,EOT, unscheduled visit
  Correlation between IMP4297 plasma concentration and QT interval
Part II: Dose Expansion safety and tolerability | From signing ICF until safety follow-up
  TEAE, vital signs, physical examinations, ECG, laboratory tests (including serum chemistry, hematology, urinalysis and coagulation), etc.
Part II: Dose Expansion anti-tumor activity | from the initiation of study drugs until documented disease progression, withdrawal of consent, loss to follow-up, death, initiation of new anti-cancer treatment or termination of study
  progression-free survival (PFS ),duration of response (DoR),Disease control rate （DCR),overall survival (OS)
Part II: Dose Expansion PK profile of IMP4297 and temozolomide | Cycle 1 Day 1,Cycle 1 Day 15,Cycle 2 Day 1,Any cycle after cycle 2,unscheduled visit
  PK parameters derived from IMP4297 and temozolomide plasma concentration data
Part II: Dose Expansion effect of IMP4297 on QT interval | Cycle 1 Day 1,Cycle 1 Day 15,Cycle 2 Day 1,CnD1,EOT, unscheduled visit
  Correlation between IMP4297 plasma concentration and QT interval

CONTACTS AND LOCATIONS:
Locations (21):
- United States (4):
  - GenHarp Clinical Solutions, Evergreen Park, Illinois
  - Gabrail Cancer Researh Center, Canton, Ohio
  - Mark H. Zangmeister Center, Columbus, Ohio
  - Sarah Cannon Research Institute - Tennessee Oncology, Tennessee City, Tennessee
- Australia (4):
  - Border Medical Oncology, Albury, New South Wales
  - Blacktown Hospital, Blacktown, New South Wales
  - Orange Hospital, Orange, New South Wales
  - Peninsula Health Frankston Hospital, Frankston, Victoria
- China (4):
  - Beijing Cancer Hospital, Beijing
  - Jilin Cancer Hospital, Jilin
  - Fudan University Shanghai Cancer Center, Shanghai
  - Hubei Cancer Hospital, Wuhan
- South Korea (4):
  - Chungbuk National University Hospital, Cheongju-si
  - The Catholic university of Korea, st. Vincent's Hospital, Gyeonggi-do
  - Yonsei university health system, Severance Hospital, Seoul
  - Asan Medical Center, Seoul
- Taiwan (5):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation Linko, Taoyuan District

IPD SHARING:
Plan to Share IPD: No